CLINICAL TRIAL: NCT07158385
Title: Impact of Dietary Protein and Fat on Postprandial Glycemic Response in Adolescents With Type 1 Diabetes and Assessment of the Management of This Response Through Insulin Regimen
Brief Title: Effect of High Fat High Protein Meal in Type 1 Diabetes
Acronym: T1DM-HFHP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Collaborators: Hacettepe University (Other)
Responsible Party: Principal Investigator, Nurcan Bağlam, Assistant Professor, Cumhuriyet University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 17-AKD-195
Record Dates: First submitted 2025-08-28; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Type 1 Diabetes Mellitus; Adolescent
Keywords: Type 1 diabetes; carbohydrate counting; fat protein counting; glycemic response
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Qa-SNARE Proteins

STUDY DESIGN:
Intervention Model Description: Four different interventions were applied to the same individuals
Masking Description: Participant blinded for insulin administration
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Clinical group (Experimental): Each participant attended all 4 test meals
  Interventions: Other: Standard test meal (SM); Other: High fat high protein meal-carbohydrate counting (HFHP); Other: High fat high protein meal-fat counting (HFHP-a); Other: High fat high protein meal-fat and protein counting (HFHP-b)

INTERVENTIONS:
Other: Standard test meal (SM) — Participants were given a standard breakfast meal with a fat and protein content similar to their daily intake. Insulin was administered according to their individual carbohydrate-to-insulin ratio. On the test day, venous blood samples were collected from the catheter inserted for GLP-1, glucagon, and free fatty acid analysis immediately before the meal (t=0 minute) and at 30, 60, 90, 120, 240, and 360 minutes after the meal.
  Other Names: Carb counting
Other: High fat high protein meal-carbohydrate counting (HFHP) — On the high-fat, high-protein meal-carbohydrate counting test day (HFHP), participants were given a high-fat and high-protein breakfast. Insulin was administered according to the individual carbohydrate-to-insulin ratio. On the test day, venous blood samples were collected from the catheter inserted for GLP-1, glucagon, and free fatty acid analysis immediately before the meal (t=0 minute) and at 30, 60, 90, 120, 240, and 360 minutes after the meal.
  Other Names: Carb counting
Other: High fat high protein meal-fat counting (HFHP-a) — On the high-fat, high-protein meal-fat-counting test day (HFHP-a), participants were given a high-fat and protein breakfast. In addition to their individual carbohydrate/insulin ratio, insulin was administered based on fat counting (1 unit for every 15 g of fat after the first 15 g of fat in the meal). In this method, the insulin dose calculated based on their individual carbohydrate/insulin ratio was delivered via insulin pump as a standard bolus, while the insulin dose calculated based on their fat count was delivered as a 4 hour extended bolus.
  Other Names: Carb and fat counting
Other: High fat high protein meal-fat and protein counting (HFHP-b) — On the high-fat, high-protein meal-fat and protein counting test day (HFHP-b), participants were given a high-fat and protein breakfast. In addition to the individual carbohydrate/insulin ratio, insulin was administered according to the adapted Pankowska Algorithm (1 FPU for every 100 kcal after the first 200 kcal of the meal). In this method, the insulin dose calculated based on the individual carbohydrate/insulin ratio was delivered as a standard bolus by an insulin pump, while the insulin dose calculated based on the fat and protein count was delivered as a spread over 4 hours.
  Other Names: Carb and fat-protein counting

SUMMARY:
Aim: Despite optimal glycemic control in individuals with type 1 diabetes, post-meal hyperglycemia remains a clinical challenge, and it has been identified as an independent risk factor for the development of long-term complications, including cardiovascular diseases. With the increasing use of continuous glucose monitoring systems, evidence has been obtained that traditional insulin dosing strategies are not sufficiently effective as the effects of meals with different macronutrient content on glycemic response are further illuminated. It is argued that relying solely on counting carbohydrates for achieving glycemic control is insufficient, and that proteins and fats can cause an increase in postprandial glycemic response. Therefore, it is necessary for Type 1 diabetics to determine insulin dosage based not only on carbohydrates, but also on the amount of fats and proteins in their meals. This study investigated the protein and fat counting in addition to carbohydrate counting on the postprandial blood glucose levels in adolescents with Type 1 diabetes and analyzed the effect of the dietary fat and protein on glucagon, glucagon-like peptide-1 (GLP-1) and free fatty acid (FFA) levels.

Methods: In this single center, randomised controlled, single-blind study with regards to insulin, 11 adolescents aged 12-18 years using continuous subcutaneous insulin infusion (CSII) were given standard meal (SM), and three test meals (HFHP: high-fat-high-protein meal using carbohydrate counting; HFHP-a: high-fat-high-protein meal using carbohydrate and fat counting; HFHP-b: high-fat-high-protein meal using carbohydrate and fat-protein counting) to compare postprandial 6 hours glucose response using continuous glucose monitoring system (CGMS). Also postprandial plasma glucagon, FFA, and GLP-1 levels were compared for 6 hours after a standard meal and a high-fat-high-protein meal.

DETAILED DESCRIPTION:
This study is designed as a single-center, randomized, controlled, single-blind study on insulin. Eleven adolescents aged 12-18 years receiving continuous subcutaneous insulin infusion (CSII) were administered a standard meal (SM) and three test meals (HFHP: high-fat-high-protein meal using carbohydrate counting; HFHP-a: high-fat-high-protein meal using carbohydrate and fat counting; HFHP-b: high-fat-high-protein meal using carbohydrate and fat-protein counting) to compare 6-hour postprandial glucose responses using continuous glucose monitoring system (CGMS). The standard meal contained 58.6 g carbohydrate, 16.9 g protein, 14.8 g fat, while the high-fat high-protein meal contained 58.2 g carbohydrate, 32.4 g protein, 30.4 g fat. CGMS were extracted from the cases and transferred to the computer, and their analysis was performed by the researcher, taking into account the capillary blood sugar measurements in the diary. Early (0-120 min), late (120-360 min), and total (0-360 min) glycemic response for the standard and test meals were analyzed using the calculation of the "incremental area under the curve" (iAUC) method. In addition, TIR (time in range) (70-180 mg/dL) and TAR (time above range) (>180 mg/dL) values obtained at early (0-120 min), late (120-360 min) and total (0-360 min) periods during the test meals of the participants were compared. Additionally, venous blood samples taken with the inserted catheter on the test day just before (t=0th min) the standard meal (SM) and high-fat high-protein meal (HFHP), and at the 30th, 60th, 90th, 120th, 240th and 360th minutes after the meal. 6-hour postprandial plasma glucagon, FFA, and GLP-1 levels were compared after the standard meal and the high-fat-high-protein meal. Early (0-120 min), late (120-360 min), and total (0-360 min) total area under the curve (tAUC) method was used to compare glucagon, GLP-1 and free fatty acid levels.

ELIGIBILITY:
Inclusion Criteria:

* No chronic disease other than type 1 diabetes mellitus
* Receiving continuous insulin infusion pump therapy

Exclusion Criteria:

* The individual's insulin requirement is less than 0.5 IU/kg/day
* High HbA1c (>8%)
* Presence of complications (Microalbuminuria, etc.)
* Presence of a comorbidity (Celiac disease, etc.)
* New initiation of CSII treatment (<6 months)
* Living outside Ankara
* Parental and individual reluctance
* The individual refuses to donate blood during the test meals

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 11 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2021-02-17 (Actual)

PRIMARY OUTCOMES:
Glucose response | For each intervention meal (4 interventions), participants' glucose response was assessed for 6 hours after the meals.
  Glucose response was measured using continuous glucose monitoring system (CGMS). CGMS were extracted from the cases and transferred to the computer, and their analysis was performed by the researcher, taking into account the capillary blood sugar measurements in the diary. Early (0-120 min), late (120-360 min), and total (0-360 min) glycemic response for the standard and test meals were analyzed using the calculation of the "incremental area under the curve" (iAUC) method. In addition, TIR (time in range) (70-180 mg/dL) and TAR (time above range) (>180 mg/dL) values obtained at early (0-120 min), late (120-360 min) and total (0-360 min) periods during the test meals of the participants were compared.
Plasma GLP-1 measurement | On the test day just before (t=0th min) the standard meal (SM) and high-fat high-protein meal (HFHP), and at the 30th, 60th, 90th, 120th, 240th and 360th minutes after the meal.
  Venous blood samples were taken from two intervention meals, a standard meal (SM) and a high-fat high-protein meal (HFHP), and were evaluated using an ELISA kit. Mean values at time points and early (0-120 min), late (120-360 min), and total (0-360 min) area under the curve (tAUC) method was used to compare the GLP-1 levels.
Plasma glucagon measurement | Venous blood samples taken with the inserted catheter on the test day just before (t=0th min) the standard meal (SM) and high-fat high-protein meal (HFHP), and at the 30th, 60th, 90th, 120th, 240th and 360th minutes after the meal.
  Venous blood samples were taken from two intervention meals, a standard meal (SM) and a high-fat high-protein meal (HFHP), and were evaluated using an ELISA kit. Mean values at time points and early (0-120 min), late (120-360 min), and total (0-360 min) area under the curve (tAUC) method was used to compare the glucagon levels.
Plasma free fatty acid measurement | On the test day just before (t=0th min) the standard meal (SM) and high-fat high-protein meal (HFHP), and at the 30th, 60th, 90th, 120th, 240th and 360th minutes after the meal.
  Venous blood samples were taken from two intervention meals, a standard meal (SM) and a high-fat high-protein meal (HFHP), and were evaluated using an ELISA kit. Mean values at time points and early (0-120 min), late (120-360 min), and total (0-360 min) area under the curve (tAUC) method was used to compare the free fatty acid levels.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Alev Özön, MD, Prof., Study Chair — Hacettepe University; Hülya Gökmen Özel, Prof. Dr., Study Director — Hacettepe University; Elmas Nazlı Gönç, MD, Prof., Principal Investigator — Hacettepe University; Ayfer Alikaşifoğlu, MD, Prof., Principal Investigator — Hacettepe University; Oytun Portakal, Assoc. Prof. Dr., Principal Investigator — Hacettepe University
Locations (1):
- Sivas Cumhuriyet University, Faculty of Health Sciences, Department of Nutrition and Dietetics, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smart CE, Evans M, O'Connell SM, McElduff P, Lopez PE, Jones TW, Davis EA, King BR. Both dietary protein and fat increase postprandial glucose excursions in children with type 1 diabetes, and the effect is additive. Diabetes Care. 2013 Dec;36(12):3897-902. doi: 10.2337/dc13-1195. Epub 2013 Oct 29. PMID 24170749